CLINICAL TRIAL: NCT03426215
Title: Observational Study on the Long-Term Course of Integrative Korean Medicine Treatment for Lumbar Intervertebral Disc Herniation: Prospective Multicenter 10 Year Follow-up
Brief Title: Long-Term Course of Korean Medicine Treatment for Lumbar Disc Herniation
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2017-13
Record Dates: First submitted 2018-02-01; First posted 2018-02-08 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Low Back Pain; Sciatica; Intervertebral Disc Displacement
MeSH Terms: conditions — Low Back Pain; Sciatica; Intervertebral Disc Displacement | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ten year follow-up group: No interventions will be administered (Magnetic Resonance Imaging (MRI) will be administered as an outcome measurement).
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) — Changes in size and severity of the main herniated disc causing radiating pain will be evaluated by radiology specialists and Korean medicine doctors (KMDs) and categorized into three groups (improved, worse or no discernible change) in comparison with the immediate previous MRI to track long-term changes and assess for correlations in subjective clinical symptoms and objective physical evaluation and MRI results.

SUMMARY:
This observational study will assess the long-term course and effect of Korean medicine treatment in lumbar intervertebral disc herniation patients who received integrative Korean medicine treatment for 24 weeks as part of a previous clinical study.

DETAILED DESCRIPTION:
This observational study will assess the long-term course and effect of Korean medicine treatment in lumbar intervertebral disc herniation patients with a main complaint of radiating leg pain who received integrative Korean medicine treatment for 24 weeks at Jaseng Hospital of Korean Medicine (Gangnam main branch) as part of a previous clinical study which was conducted from November, 2006 to April, 2007, and give written informed consent to long-term follow-up assessment at 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar intervertebral disc herniation patients with a main complaint of radiating leg pain who received integrative Korean medicine treatment for 24 weeks at Jaseng Hospital of Korean Medicine (Gangnam main branch) as part of a previous clinical study which was conducted from November, 2006 to April, 2007
* Patients who give voluntary written informed consent to long-term follow-up assessment (quantitative and qualitative questionnaires, and MRI) at 10 years.

Exclusion Criteria:

* Patients who cannot give voluntary written informed consent to this study or answer study questionnaires (e.g. severe psychological disorders)
* Patients participating in other clinical studies or otherwise deemed unsuitable by the researchers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lumbar intervertebral disc herniation patients with a main complaint of radiating leg pain who received integrative Korean medicine treatment for 24 weeks at Jaseng Hospital of Korean Medicine (Gangnam main branch) as part of a previous clinical study which was conducted from November, 2006 to April, 2007.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2018-04-28 (Actual); Study Completion 2018-04-28 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analogue Scale (VAS) of radiating leg pain | Difference from baseline at 10 years
  Visual Analogue Scale (VAS) uses a 10cm line labeled at each end with scale anchors. In pain measurement using VAS, patients are asked to mark a point that represents their pain between the anchors of 'no pain (minimum score: 0)' and 'worst pain imaginable (maximum score: 100)'. Total scores are recorded in millimeters with a total range of 0-100 millimeters. Higher VAS values represent more severe pain, and a greater change from baseline (If baseline - follow up is a positive value) indicates a better outcome.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) of low back pain | Baseline, and 10 years
  Visual Analogue Scale (VAS) uses a 10cm line labeled at each end with scale anchors. In pain measurement using VAS, patients are asked to mark a point that represents their pain between the anchors of 'no pain (minimum score: 0)' and 'worst pain imaginable (maximum score: 100)'. Total scores are recorded in millimeters with a total range of 0-100 millimeters. Higher VAS values represent more severe pain.
Visual Analogue Scale (VAS) of radiating leg pain | Baseline, and 10 years
  Visual Analogue Scale (VAS) uses a 10cm line labeled at each end with scale anchors. In pain measurement using VAS, patients are asked to mark a point that represents their pain between the anchors of 'no pain (minimum score: 0)' and 'worst pain imaginable (maximum score: 100)'. Total scores are recorded in millimeters with a total range of 0-100 millimeters. Higher VAS values represent more severe pain.
Numeric Rating Scale (NRS) of low back pain | Baseline, and 10 years
  In pain measurement using Numeric Rating Scale (NRS), patients are asked to rate their pain by selecting a number from 0 to 10 that best represents their pain severity between the anchors of 0 which indicates 'no pain', and 10 which indicates 'worst pain possible'.
Numeric Rating Scale (NRS) of radiating leg pain | Baseline, and 10 years
  In pain measurement using Numeric Rating Scale (NRS), patients are asked to rate their pain by selecting a number from 0 to 10 that best represents their pain severity between the anchors of 0 (minimum score) which indicates 'no pain', and 10 (maximum score) which indicates 'worst pain possible'. Higher NRS values represent more severe pain.
Oswestry Disability Index (ODI) | Baseline, 10 years
  The ODI is a 10-item questionnaire developed to assess level of disability due to low back pain (LBP). Each item is graded into 6 levels, each representing a score of 0-5. Higher scores indicate greater limitation relating to LBP.
36-Item Short Form Survey (SF-36) | Baseline, 10 years
  SF-36 consists of 36 items across 8 domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. SF-36 is used to rate functional health and well-being in patients and healthy individuals. Higher scores indicate better HRQoL.
Patient Global Impression of Change (PGIC) | Baseline, 10 years
  PGIC grades the level of subjective improvement into 7 levels (1, very much improved; 2, much improved; 3, slightly improved; 4, no change; 5, slightly worse; 6, much worse; and 7, very much worse).
Lumbar range of movement (ROM) | Baseline, 10 years
  ROM measurements are valid (r=0.97) and reliable (r=0.94), but not highly responsive (effect size=0.1-0.6). If ROM is uncheckable from pain, the angle will be recorded as 0°.
Straight leg raise (SLR) test | Baseline, 10 years
  While SLR measurements are reliable (intraclass correlation coefficient=0.95), they are not very responsive (effect size=0.2). If SLR is uncheckable from pain, the angle will be recorded as 0°.
Qualitative questionnaire on 10 year course | 10 years
  The qualitative questionnaire on 10 year course and outcome since receiving integrative Korean medicine treatment used in this study is a 14-item descriptive evaluation encompassing various items (a mixture of short-answer questions, multiple choices, and transcript of essay form answers) on the change before and after treatment over the course of 10 years (e.g. change in perception of surgery and non-surgical treatment, change in everyday life or habits, and treatment recommendation to others).
Medical history | 10 years
  Physicians will rate the causal relationship of each treatment from the previous clinical study with the patient's medical history potentially associated with treatment on a 6-point scale (1, definitely related; 2, probably related; 3, possibly related; 4, probably not related; 5, definitely not related; and 6, unknown), and classify all medical history potentially associated with treatment with the Spilker classification, which has 3 grades (1, mild: no intervention needed and does not greatly impede normal activity (function) of patient; 2, moderate: significantly impedes normal activity (function) of patient, and may need intervention, with subsequent resolution; 3, severe: severe adverse event needing intensive intervention, leaving sequela).
Adverse events | 10 years
  Adverse events potentially associated with MRI will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Me-riong Kim, KMD, M.Sc., Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No